CLINICAL TRIAL: NCT05416788
Title: Effect of Cervical Manipulation on Mouth Opening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Americas (Other)
Responsible Party: Principal Investigator, Ignacio Astudillo Ganora, principal investigator, University of Americas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60/2022
Record Dates: First submitted 2022-06-06; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Bruxism; Face Pain
MeSH Terms: conditions — Bruxism; Facial Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical manipulation group (Experimental): high-velocity, low-amplitude cervical manipulation
  Interventions: Other: cervical manipulation
- Control group (Sham Comparator): placebo manipulation, the cervical spine will be tilted and rotated without reaching the end feel or the pump
  Interventions: Other: Sham intervention

INTERVENTIONS:
Other: cervical manipulation — high-velocity, low-amplitude cervical manipulation
  Arms: Cervical manipulation group
Other: Sham intervention — lateral flexion and cervical rotation without manipulation
  Arms: Control group

SUMMARY:
Objectives: To compare the effects of cervical manipulation on the ranges of motion of

mouth opening and painful pressure points in the masseter and temporal muscles after

of cervical manipulation compared to the control group.

Material and methods: Single-blind randomized clinical trial with two arms, one group

intervention and a control group.

Hypothesis: There is a significant difference in mouth opening and painful pressure points

between the intervention group and the control group.

Expected results: The intervention group would significantly increase their mouth opening

maximal and decrease pressure pain in the masseter and temporalis muscles.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years of age, men and women
* Students with neck and/or facial pain minimum 3/10 VAS scale
* Kinesiology students who regularly attend face-to-face classes

who have a mobility pass and a health declaration.

· Students who read and sign the informed consent.

Exclusion Criteria:

* Orthognathic surgery
* Head and neck fracture or injury
* Contraindication (red flag) to perform high-speed, low-amplitude cervical manipulation (bone cancer, osteoporosis, vertebral artery injury, etc.)
* Positive cervical safety tests (example: Klein test positive)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
normal mouth opening in millimeters | Change from Baseline mouth open at 5 minutes
  With a buccal goniometer, the maximum mouth opening will be measured in millimeters.

SECONDARY OUTCOMES:
masseter muscle pressure points | Change from Baseline pain points at 5 minutes
  Pain points will be measured under pressure with a pressure pain meter or algo meter. This measurement will be measured in kilograms.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de las Americas, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No